CLINICAL TRIAL: NCT02624739
Title: Initial Assessment of the Usability of Remote Monitoring of Respiration Parameters in the Routine Management of Heart Failure Patients
Brief Title: Reassure Remote Respiration Monitoring in Heart Failure Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for study was withdrawn.
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AGH-11-15-01
Record Dates: First submitted 2015-11-20; First posted 2015-12-08 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: respiration rate, sleep
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Reassure Non-Contact Respiration Monitor: Respiration parameters transmitted by the Reassure device will be evaluated daily by the study team and participants will be contacted for further evaluation if a change in respiration patterns is noted. Participants will continue with standard of care heart failure treatment.
  Interventions: Device: Reassure Non-Contact Respiration Monitor
- Control (Active Comparator): Reassure Non-Contact Respiration Monitor: Respiration parameters will be transmitted and stored, but there will be no active evaluation of respiration patterns. Participants will continue with standard of care heart failure treatment.
  Interventions: Device: Reassure Non-Contact Respiration Monitor

INTERVENTIONS:
Device: Reassure Non-Contact Respiration Monitor — Reassure uses a specially-designed, non-contact motion sensor to monitor body movement and continuous respiratory rate (CRR) during sleep. Reassure is used to monitor, over a prolonged period, the sleep patterns and respiration rate while the patient is asleep.

SUMMARY:
This study is designed to descriptively assess improvement in quality of life and test the usability of remotely monitored respiration parameters in the routine management of recently discharged heart failure patients. It will consist of two arms: (i) intervention, and (ii) control. Participants will be randomized to either arm at time of enrollment. Every participant enrolled in the study will receive a device for remote monitoring.

DETAILED DESCRIPTION:
Heart failure ('HF') presents an increasing social and economic burden, especially with respect to HF related hospitalizations. Some commentators suggest that these costs may double within the next two decades. Respiration patterns are well acknowledged as having diagnostic and prognostic value in HF. In this preliminary study, the investigators assess the usability of remote monitoring of respiration parameters in the routine management of HF patients.

Objectives: (primary and important secondary objectives)

The primary aims are:

1. Assess usability of the system (primary measurement is % of successful data transmissions from participants' homes, secondary measurement includes scores from the System Usability Scale)
2. Assess quality of life (as measured using the KCCQ) for HF patients monitored with a non-contact respiration monitor which can be used by clinicians to guide standard therapy.

Other key secondary objectives include examining trends in healthcare utilization, descriptively assessing any differences in care patterns post hoc between participants.

As part of the study plan , the investigators will also analyze respiration and sleeping patterns from the raw data files to assess the prevalence of unusual breathing patterns such as sleep apnea in newly discharged HF patients and how these patterns may be linked to outcomes. These analyses will be executed retrospectively on a population rather than individual participant basis and will not be used to inform individual treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥18 years old
* Patients admitted to hospital for worsening of heart failure; Worsening of heart failure is defined as symptoms consistent with worsening of heart failure, including dyspnea and an elevated BNP. Patients must have existing diagnosis of heart failure, either preserved ejection fraction or reduced ejection fraction (HFpEF or HFrEF)
* Weight ≥35 kg
* Pre-Menopausal Women ≥18 years of age must have a negative urine/serum pregnancy test or pre-menopausal women with evidence of surgical sterilization or post-menopausal women.
* Must qualify for standard home care post discharge
* Must be able to read and understand English and consent for themselves

Exclusion Criteria:

* Under 18 years of age
* Participant is on a form of non-invasive positive airway pressure ventilation (in such cases, respiratory rates and variability will reflect combined physiology plus machine effect)
* Participant has an existing diagnosis in the medical record for sleep disordered breathing, whether on therapy or not
* Participant has cognitive impairment (determined by physician) that will make it hard for them to follow instructions regarding therapy usage
* BMI> 40
* Patients who are discharged to hospice care, Skilled Nursing Facilities or Long Term Acute Care facilities
* Patients who are actively being monitored using a pulmonary arterial pressure monitor (CardioMEMs)
* Patients with COPD GOLD Stage III or IV
* Planned procedures at time of discharge that will occur within timeframe of study that will require hospitalization etc.
* Participant declines to participate at any time.
* Patients involved in therapy intervention clinical trials
* Any investigational drug use within 30 days prior to enrollment.
* Pregnant or lactating females.
* Participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures
* Participants who have no cellular coverage at their primary residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06-02 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Patarroyo-Aponte, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated after enrollment but prior to data collection
Period: Overall Study
Arm/Group | Intervention | Control
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated after enrollment but prior to data collection
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Percent Successful Data Transmissions
Description: Number of successful data transmissions compared to number of possible data transmissions
Time Frame: One year
Population: Study terminated prior to enrollment
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Quality of Life as Measured by Kansas City Cardiomyopathy Questionnaire
Description: Quality of life as measured by Kansas City Cardiomyopathy Questionnaire
Time Frame: One year
Population: study terminated prior to enrollment
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: System Usability
Description: Usability of the system by the clinical care team as measured by a System Usability Scale
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Healthcare Utilization
Description: Trends in healthcare utilization and care patterns as measured by numbers of home visits, outpatient visits, all-cause hospitalizations, HF related hospitalizations, lengths of stay
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: HF Drug Compliance
Description: Percent compliance in HF-specific drugs: diuretics, ACE/ARB, Beta Blockers, Spironolactone/Nitrates and Hydralazine
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: HF Drug Changes
Description: Rate of changes in HF-specific drugs: diuretics, ACE/ARB, Beta Blockers, Spironolactone/Nitrates and Hydralazine
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Biomarkers
Description: Trends in HF-specific biomarkers: NT-proBNP, ST2
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Respiration Patterns
Description: Retrospective exploratory analysis of respiration rate measured by the Reassure device compared to participant outcomes (eg, status at end of study, changes in medications, biomarkers, etc) to evaluate potential predictive trends for use in designing future studies.
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Sleeping Patterns
Description: Retrospective exploratory analysis of sleeping patterns measured by the Reassure device compared to participant outcomes (eg, status at end of study, changes in medications, biomarkers, etc) to evaluate potential predictive trends for use in designing future studies.
Time Frame: One year
Population: study terminated
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated after enrollment but prior to data collection
Description: The study was terminated after enrollment but prior to data collection
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No